CLINICAL TRIAL: NCT00306644
Title: Effect of Rosiglitazone and Placebo on Carotid Intima Media Thickness in Patients With Insulin Resistance Syndrome and/or Type 2 Diabetes
Brief Title: Effect Of Rosiglitazone On Carotid Intima Media Thickness In Patients With Insulin Resistance Syndrome And/Or Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49653/334
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: rosiglitazone; Type 2 diabetes; intima media thickness; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm 1 (Experimental): study drug
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — study drug

SUMMARY:
The study investigated the effect of rosiglitazone and placebo on carotid intima media thickness in patients with insulin resistance syndrome and/or type 2 diabetes.

DETAILED DESCRIPTION:
RAS Rosiglitazone and Atherosclerosis Study: A 1 year randomised, double-blind, parallel group, placebo controlled study to evaluate the efficacy of rosiglitazone on the progression of intima-media thickness in the carotid artery in subjects with insulin resistance syndrome and/or type 2 diabetes mellitus

ELIGIBILITY:
Inclusion criteria:

* insulin resistant syndrome or Type 2 Diabetes.

Exclusion criteria:

* Use of >= 2 concomitant oral antihyperglycaemic agents within 3 months of study start.
* Initiation of anti-hypertensive or lipid lowering therapy <= 6 months prior to study start or who increased the dose 3 months prior to study start.
* Unstable or severe angina or congestive heart failure NYHA class i-iv, history of acute myocardial infarction or stroke within last 6 months.
* Any history of surgical intervention in the right carotid artery.
* Clinically significant hepatic disease.
* Creatinine clearance <40ml/min.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2002-05; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the composite intima-media thickness (IMT) in the carotid artery following 52 weeks of treatment. | 52 weeks

SECONDARY OUTCOMES:
Plaque occurrence & stenosis within the right carotid artery. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Hedblad B, Zambanini A, Nilsson P, Janzon L, Berglund G. Rosiglitazone and carotid IMT progression rate in a mixed cohort of patients with type 2 diabetes and the insulin resistance syndrome: main results from the Rosiglitazone Atherosclerosis Study. J Intern Med. 2007 Mar;261(3):293-305. doi: 10.1111/j.1365-2796.2007.01767.x. PMID 17305652
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 49653/334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 49653/334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 49653/334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 49653/334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 49653/334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 49653/334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 49653/334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register